CLINICAL TRIAL: NCT02962531
Title: A Randomized, Single-Dose, 3-Way Crossover Study to Evaluate the Relative Bioavailability of the IX-01 Caplet Formulation Compared With the IX 01 Aqueous Dispersion Formulation, and the Effect of Food on the IX-01 Caplet Formulation, in Healthy Male Subjects
Brief Title: Relative Bioavailability Study of IX-01 Caplet Versus Aqueous Dispersion and Food Effect of the Caplet in Healthy Males
Acronym: IX-0106 RBA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ixchelsis Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IX-0106
Record Dates: First submitted 2016-10-24; First posted 2016-11-11 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): A single 1600 mg (4 x 400 caplets) oral dose of IX-01 under fasted conditions
  Interventions: Drug: IX-01 caplets 1600 mg (4 x 400 mg), fasted
- Treatment B (Experimental): A single 1600 mg (4 x 400 caplets) oral dose of IX-01 under fed conditions
  Interventions: Drug: IX-01 caplets 1600 mg (4 x 400 mg), fed
- Treatment C (Experimental): A single 1600 mg aqueous dispersion (20 mL) oral dose of IX-01 under fasted conditions.
  Interventions: Drug: IX-01 aqueous dispersion 1600 mg (20 mL), fasted

INTERVENTIONS:
Drug: IX-01 caplets 1600 mg (4 x 400 mg), fasted — oral dose under fasted conditions
  Arms: Treatment A
Drug: IX-01 caplets 1600 mg (4 x 400 mg), fed — oral dose under fed conditions
  Arms: Treatment B
Drug: IX-01 aqueous dispersion 1600 mg (20 mL), fasted — oral dose under fasted conditions
  Arms: Treatment C

SUMMARY:
An open-label, randomized, three-period, three-way crossover trial of single doses of IX-01 in 12 healthy male subjects. In each period, subjects will receive a single oral dose of 1600 mg IX-01, either as an aqueous dispersion in a fasted state, or as caplets in the fed or fasted state

DETAILED DESCRIPTION:
This is a Relative Bioavailability Study to compare single oral doses of 1600mg IX-01, either as an aqueous dispersion in a fasted state, or as caplets in the fed or fasted state. Each volunteer in the study will receive each of the formulations listed below. Each formulation will be separated by at least a 5-day drug-free (washout) period.

* Treatment A: A single 1600 mg (4 x 400 caplets) oral dose of IX-01 under fasted conditions
* Treatment B: A single 1600 mg (4 x 400 caplets) oral dose of IX-01 under fed conditions
* Treatment C: A single 1600 mg aqueous dispersion (20 mL) oral dose of IX-01 under fasted conditions.

In the fasted treatment periods, dosing will follow an overnight fast of at least 10 hours.

In the fed treatment period, following an overnight fast of at least 10 hours, a standard high-calorie, high-fat breakfast meal will be given 30 minutes prior to administration of the study drug.

There will be a final follow-up visit 7-10 days after the final dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 30 kg/m2
* Body weight of ˃60 kg (132 lbs) at screening
* Able to understand the nature of the trial and any hazards of participating. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of the entire trial
* Willing to comply with the contraception requirements of the trial
* Willing to give written consent to participate
* Willing and able to remain in the study unit for the entire duration of each confinement period and return for outpatient visits
* Willing and able to consume the entire high-calorie, high-fat breakfast meal in the designated timeframe required during fed study period
* Vital signs at both screening and at baseline within: heart rate: 50-90 beats per minute; systolic blood pressure: 100-130 mmHg; diastolic: 60-90 mmHg

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at screening that could interfere with the objectives of the trial or safety of the volunteer, including any of the following:
* Lipid and/or liver function test results >1.25 times upper limit of normal or another clinical laboratory result judged clinically significant
* An international normalised ratio of >1.2 or a platelet count <150 x10^3/mL
* History of unexplained syncope
* Family history of unexplained sudden death or sudden death due to long QT syndrome
* QTcF interval >450 msec at screening
* Bundle branch block or another conduction abnormality during an ECG, other than mild first degree atrio-ventricular block, judged clinically significant
* Irregular rhythms during an ECG, other than sinus arrhythmia or occasional supraventricular ectopic beats, judged clinically significant
* T-wave configuration of insufficient quality for determination of QT interval, as assessed by ECG and judged clinically significant by the Investigator
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate participation in the trial or make study participation unnecessarily hazardous
* Impaired gastrointestinal, endocrine, thyroid, hepatic, cardiovascular, respiratory, hematological, renal or neurological function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness
* Surgery (e.g. stomach bypass) or medical condition that might affect absorption, metabolism, or elimination of medicines
* Presence or history of severe adverse reaction to any drug and/or a history of skin reactions (rashes) to any drug
* Previous allergic response which involved hives, swelling, shortness of breath, or anaphylaxis
* Has used any over-the-counter medications, nutritional or dietary supplements, herbal preparations, or vitamins, except short courses of medication (such as acetaminophen), that could interfere with subject safety or the integrity of the trial data within 7 days prior to the first dose of medication
* Any prescription medication within 14 days prior to the first dose of study medication
* Participation in another clinical trial within 60 days prior to the first dose of study medication
* Previous participation in this trial or any other clinical trial of an oxytocin receptor antagonist
* Presence or history of drug or alcohol abuse, or intake of more than 21 units of alcohol weekly or more than 5 cigarettes daily
* Unwilling or unable to comply with all protocol requirements
* Positive urine screen for drugs of abuse
* Positive for hepatitis B surface antigen, hepatitis C antibody or Human Immunodeficiency Virus at screening or previously treated for hepatitis B, hepatitis C, or Human Immunodeficiency Virus infection
* Donated blood or plasma within 30 days prior to the first dose of study medication
* Employee of the investigator site or any company involved in sponsoring, organizing, or conducting the trial, or immediate family of the employee

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter peak plasma concentration of IX-01 (C max) | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  Relative bioavailability of the caplet formulation of IX-01compared with the aqueous dispersion formulation when administered in the fasted state
Pharmacokinetic parameter time of peak plasma concentration of IX-01 (t max) | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  Relative bioavailability of the caplet formulation of IX-01compared with the aqueous dispersion formulation when administered in the fasted state
Pharmacokinetic parameter terminal half-life (t 1/2) | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  Relative bioavailability of the caplet formulation of IX-01compared with the aqueous dispersion formulation when administered in the fasted state
Pharmacokinetic parameter elimination rate constant (K el) | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  Relative bioavailability of the caplet formulation of IX-01compared with the aqueous dispersion formulation when administered in the fasted state
Relative bioavailability of the caplet formulation of IX-01 compared with the aqueous dispersion formulation (fasted) | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  Relative bioavailability of the caplet formulation of IX-01compared with the aqueous dispersion formulation when administered in the fasted state
Pharmacokinetic parameter area under the concentration-time curve (AUC 0-inf) | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  Relative bioavailability of the caplet formulation of IX-01compared with the aqueous dispersion formulation when administered in the fasted state
area under the concentration-time curve from 0 up to the time of last quantifiable concentration (AUC last) | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  Relative bioavailability of the caplet formulation of IX-01compared with the aqueous dispersion formulation when administered in the fasted state
The relative bioavailability of IX-01, as judged by AUC 0-inf (F rel) | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  Relative bioavailability of the caplet formulation of IX-01 compared with the aqueous dispersion formulation when administered in the fasted state
Comparison of Maximum Plasma Concentration [Cmax] in fed versus fasted states | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  To determine the effect of a high-fat meal on the pharmacokinetic profile of the IX-01 caplet formulation
Comparison of Area Under the Curve [AUC] in fed versus fasted states | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  To determine the effect of a high-fat meal on the pharmacokinetic profile of the IX-01 caplet formulation
Comparison of Time to Maximum Plasma Concentration [Tmax] in fed versus fasted states | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  To determine the effect of a high-fat meal on the pharmacokinetic profile of the IX-01 caplet formulation
Comparison of the Area Under the Curve [AUC] in fed versus fasted states | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
  To determine the effect of a high-fat meal on the pharmacokinetic profile of the IX-01 caplet formulation

SECONDARY OUTCOMES:
Safety monitoring - adverse events, laboratory data, ECGs, vital signs | Day 0 to Day 21
  To monitor the safety and tolerability of IX-01

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials Early Phase Services, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No